CLINICAL TRIAL: NCT02605135
Title: Host Response to Pessaries in Microbial Communities of the Postmenopausal
Brief Title: Host Response to Pessaries in Microbial Communities of the Postmenopausal Vagina
Status: Completed | Type: Observational
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Cynthia Brincat, M.D., Ph.D., Loyola University
Other Study IDs: 207001
Record Dates: First submitted 2015-11-12; First posted 2015-11-16 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Stress Urinary Incontinence; Prolapse
MeSH Terms: conditions — Urinary Incontinence, Stress; Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Testing will consists of a vaginal swab (AIM 1) and 10 mL of vaginal lavage at each study visit.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Continued Pessary Use: All participants will undergo clinical testing prior to placement of the pessary and the investigator will test their vaginal environment prior to pessary placement. Testing will consists of a vaginal swab and 10 mL of vaginal lavage at each study visit. The participant will then be followed, and repeat testing obtained at the standard clinical interval for pessary follow-up, every three months
  Interventions: Device: Continued Pessary Use
- Discontinued Pessary Use: All participants will undergo clinical testing prior to placement of the pessary and the investigator will test their vaginal environment prior to pessary placement. Testing will consists of a vaginal swab (AIM 1) and 10 mL of vaginal lavage (Aim 2) at each study visit. The participant will then be followed, and repeat testing obtained at the standard clinical interval for pessary follow-up, every three months. Should the participant discontinue pessary use, we will additionally culture the microbes that are present on the pessary and compare those to the vaginal microbiota.
  Interventions: Device: Continued Pessary Use

INTERVENTIONS:
Device: Continued Pessary Use — Pessary Fitting

SUMMARY:
The ability to determine the postmenopausal vaginal environment and the impact of pessary use could help to maximize pessary therapy and non-surgical treatment for such a prevalent problem.

DETAILED DESCRIPTION:
The study will advance the care of elderly patients through providing data to maximize non-surgical options to those at high risk for having surgery and its attending morbidity. In characterizing substantive differences in the vaginal environment of successful and unsuccessful pessary users, the investigators can identify elderly patients at higher risk of adverse events with pessary use as well as novel targets for the pharmacologic treatment of the altered vaginal microbiota and endogenous AMP levels, potentially allowing patients to continue with non-surgical therapies rather than pursuing surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* must be English speaking
* appropriate for pessary treatment
* pelvic floor conditions such as POP (with or without the presence of a uterus), stress urinary incontinence, urge urinary incontinence, or any combination of the above.

Exclusion Criteria:

* a history of current, symptomatic vaginal stricture
* a history of current, radiation therapy,
* or current treatment with auto-immune suppression agents.
* if they have eroded mesh in the vagina from prior pelvic floor surgery

Min Age: 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects must be female, postmenopausal, and have symptomatic pelvic floor disorders as evidenced by presenting to our tertiary care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2016-04; Primary Completion 2017-11 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Predominant vaginal microorganisms of older women with and without a pessary | Baseline
  The investigator will collect a vaginal swab specimen in an aerobic and anaerobic preservative tube. Specimens will be sent to the clinical microbiology lab for quantitative culture. Expanded quantitative vaginal culture techniques and matrix assisted laser desorption ionization-time of flight mass spectrometry (MALDI-TOF MS).

SECONDARY OUTCOMES:
Vaginal antimicrobial peptide (AMP) profile of older women with and without a pessary. | Baseline
  The investigator will collect vaginal lavage fluid (VLF) prior to pessary placement and after vaginal swabs are obtained. Assessing AMP activity using high pressure liquid chromatography fractionation and radial diffusion assay to assess for AMP activity and abundance of candidate AMPs (cathelicidin, beta defensisn (hBD1 and hBD2) psoriasin, lactoferrin).
Vaginal microbiome and AMP profile between those women that choose to continue pessary use and those that do not by correlating the data from Aim 1 and Aim 2 with the clinical characteristic of continued pessary use. | 3 month visit, 6 month visit
  The investigator will collect vaginal swabs and the Vaginal Lavage Fluid for those subjects who decide to NOT have their pessaries replaced by correlating the data from outcome 1 and outcome 2 with the clinical characteristic of continued pessary use.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Brincat, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nygaard I, Barber MD, Burgio KL, Kenton K, Meikle S, Schaffer J, Spino C, Whitehead WE, Wu J, Brody DJ; Pelvic Floor Disorders Network. Prevalence of symptomatic pelvic floor disorders in US women. JAMA. 2008 Sep 17;300(11):1311-6. doi: 10.1001/jama.300.11.1311. PMID 18799443
- [Background] Hunskaar S, Burgio K, Diokno A, Herzog AR, Hjalmas K, Lapitan MC. Epidemiology and natural history of urinary incontinence in women. Urology. 2003 Oct;62(4 Suppl 1):16-23. doi: 10.1016/s0090-4295(03)00755-6. PMID 14550833
- [Background] Hendrix SL, Clark A, Nygaard I, Aragaki A, Barnabei V, McTiernan A. Pelvic organ prolapse in the Women's Health Initiative: gravity and gravidity. Am J Obstet Gynecol. 2002 Jun;186(6):1160-6. doi: 10.1067/mob.2002.123819. PMID 12066091
- [Background] Mant J, Painter R, Vessey M. Epidemiology of genital prolapse: observations from the Oxford Family Planning Association Study. Br J Obstet Gynaecol. 1997 May;104(5):579-85. doi: 10.1111/j.1471-0528.1997.tb11536.x. PMID 9166201
- [Background] Wu JM, Hundley AF, Fulton RG, Myers ER. Forecasting the prevalence of pelvic floor disorders in U.S. Women: 2010 to 2050. Obstet Gynecol. 2009 Dec;114(6):1278-1283. doi: 10.1097/AOG.0b013e3181c2ce96. PMID 19935030
- [Background] Brown JS, Waetjen LE, Subak LL, Thom DH, Van den Eeden S, Vittinghoff E. Pelvic organ prolapse surgery in the United States, 1997. Am J Obstet Gynecol. 2002 Apr;186(4):712-6. doi: 10.1067/mob.2002.121897. PMID 11967496
- [Background] Wu JM, Matthews CA, Conover MM, Pate V, Jonsson Funk M. Lifetime risk of stress urinary incontinence or pelvic organ prolapse surgery. Obstet Gynecol. 2014 Jun;123(6):1201-1206. doi: 10.1097/AOG.0000000000000286. PMID 24807341
- [Background] Smith FJ, Holman CD, Moorin RE, Tsokos N. Lifetime risk of undergoing surgery for pelvic organ prolapse. Obstet Gynecol. 2010 Nov;116(5):1096-100. doi: 10.1097/AOG.0b013e3181f73729. PMID 20966694
- [Background] Sung VW, Weitzen S, Sokol ER, Rardin CR, Myers DL. Effect of patient age on increasing morbidity and mortality following urogynecologic surgery. Am J Obstet Gynecol. 2006 May;194(5):1411-7. doi: 10.1016/j.ajog.2006.01.050. PMID 16647926
- [Background] Cundiff GW, Weidner AC, Visco AG, Bump RC, Addison WA. A survey of pessary use by members of the American urogynecologic society. Obstet Gynecol. 2000 Jun;95(6 Pt 1):931-5. doi: 10.1016/s0029-7844(00)00788-2. PMID 10831995
- [Background] Aroutcheva A, Gariti D, Simon M, Shott S, Faro J, Simoes JA, Gurguis A, Faro S. Defense factors of vaginal lactobacilli. Am J Obstet Gynecol. 2001 Aug;185(2):375-9. doi: 10.1067/mob.2001.115867. PMID 11518895
- [Background] Brotman RM, Shardell MD, Gajer P, Fadrosh D, Chang K, Silver MI, Viscidi RP, Burke AE, Ravel J, Gravitt PE. Association between the vaginal microbiota, menopause status, and signs of vulvovaginal atrophy. Menopause. 2014 May;21(5):450-8. doi: 10.1097/GME.0b013e3182a4690b. PMID 24080849
- [Background] Brotman RM, Klebanoff MA, Nansel TR, Yu KF, Andrews WW, Zhang J, Schwebke JR. Bacterial vaginosis assessed by gram stain and diminished colonization resistance to incident gonococcal, chlamydial, and trichomonal genital infection. J Infect Dis. 2010 Dec 15;202(12):1907-15. doi: 10.1086/657320. Epub 2010 Nov 10. PMID 21067371
- [Background] Hummelen R, Macklaim JM, Bisanz JE, Hammond JA, McMillan A, Vongsa R, Koenig D, Gloor GB, Reid G. Vaginal microbiome and epithelial gene array in post-menopausal women with moderate to severe dryness. PLoS One. 2011;6(11):e26602. doi: 10.1371/journal.pone.0026602. Epub 2011 Nov 2. PMID 22073175
- [Background] Nizet V, Gallo RL. Cathelicidins and innate defense against invasive bacterial infection. Scand J Infect Dis. 2003;35(9):670-6. doi: 10.1080/00365540310015629. PMID 14620153
- [Background] Luthje P, Brauner H, Ramos NL, Ovregaard A, Glaser R, Hirschberg AL, Aspenstrom P, Brauner A. Estrogen supports urothelial defense mechanisms. Sci Transl Med. 2013 Jun 19;5(190):190ra80. doi: 10.1126/scitranslmed.3005574. PMID 23785036
- [Background] Hilt EE, McKinley K, Pearce MM, Rosenfeld AB, Zilliox MJ, Mueller ER, Brubaker L, Gai X, Wolfe AJ, Schreckenberger PC. Urine is not sterile: use of enhanced urine culture techniques to detect resident bacterial flora in the adult female bladder. J Clin Microbiol. 2014 Mar;52(3):871-6. doi: 10.1128/JCM.02876-13. Epub 2013 Dec 26. PMID 24371246
- [Background] Wolfe AJ, Toh E, Shibata N, Rong R, Kenton K, Fitzgerald M, Mueller ER, Schreckenberger P, Dong Q, Nelson DE, Brubaker L. Evidence of uncultivated bacteria in the adult female bladder. J Clin Microbiol. 2012 Apr;50(4):1376-83. doi: 10.1128/JCM.05852-11. Epub 2012 Jan 25. PMID 22278835
- [Background] Collins S, Beigi R, Mellen C, O'Sullivan D, Tulikangas P. The effect of pessaries on the vaginal microenvironment. Am J Obstet Gynecol. 2015 Jan;212(1):60.e1-6. doi: 10.1016/j.ajog.2014.07.024. Epub 2014 Jul 18. PMID 25046810
- [Background] Spear GT, Zariffard MR, Cohen MH, Sha BE. Vaginal IL-8 levels are positively associated with Candida albicans and inversely with lactobacilli in HIV-infected women. J Reprod Immunol. 2008 Jun;78(1):76-9. doi: 10.1016/j.jri.2007.11.001. Epub 2008 Feb 19. PMID 18243333
- [Background] Valore EV, Wiley DJ, Ganz T. Reversible deficiency of antimicrobial polypeptides in bacterial vaginosis. Infect Immun. 2006 Oct;74(10):5693-702. doi: 10.1128/IAI.00524-06. PMID 16988245
- [Background] Mildner M, Stichenwirth M, Abtin A, Eckhart L, Sam C, Glaser R, Schroder JM, Gmeiner R, Mlitz V, Pammer J, Geusau A, Tschachler E. Psoriasin (S100A7) is a major Escherichia coli-cidal factor of the female genital tract. Mucosal Immunol. 2010 Nov;3(6):602-9. doi: 10.1038/mi.2010.37. Epub 2010 Jun 23. PMID 20571488
- [Background] Cohen MS, Britigan BE, French M, Bean K. Preliminary observations on lactoferrin secretion in human vaginal mucus: variation during the menstrual cycle, evidence of hormonal regulation, and implications for infection with Neisseria gonorrhoeae. Am J Obstet Gynecol. 1987 Nov;157(5):1122-5. doi: 10.1016/s0002-9378(87)80274-0. PMID 3120589
- [Background] Han JH, Kim MS, Lee MY, Kim TH, Lee MK, Kim HR, Myung SC. Modulation of human beta-defensin-2 expression by 17beta-estradiol and progesterone in vaginal epithelial cells. Cytokine. 2010 Feb;49(2):209-14. doi: 10.1016/j.cyto.2009.09.005. Epub 2009 Oct 9. PMID 19819163
- [Background] Frew L, Makieva S, McKinlay AT, McHugh BJ, Doust A, Norman JE, Davidson DJ, Stock SJ. Human cathelicidin production by the cervix. PLoS One. 2014 Aug 4;9(8):e103434. doi: 10.1371/journal.pone.0103434. eCollection 2014. PMID 25089904
- [Background] Radek KA, Lopez-Garcia B, Hupe M, Niesman IR, Elias PM, Taupenot L, Mahata SK, O'Connor DT, Gallo RL. The neuroendocrine peptide catestatin is a cutaneous antimicrobial and induced in the skin after injury. J Invest Dermatol. 2008 Jun;128(6):1525-34. doi: 10.1038/sj.jid.5701225. Epub 2008 Jan 10. PMID 18185531
- [Background] Barber MD, Kuchibhatla MN, Pieper CF, Bump RC. Psychometric evaluation of 2 comprehensive condition-specific quality of life instruments for women with pelvic floor disorders. Am J Obstet Gynecol. 2001 Dec;185(6):1388-95. doi: 10.1067/mob.2001.118659. PMID 11744914
- [Background] Jenkinson C, Layte R, Jenkinson D, Lawrence K, Petersen S, Paice C, Stradling J. A shorter form health survey: can the SF-12 replicate results from the SF-36 in longitudinal studies? J Public Health Med. 1997 Jun;19(2):179-86. doi: 10.1093/oxfordjournals.pubmed.a024606. PMID 9243433
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] Bump RC, Mattiasson A, Bo K, Brubaker LP, DeLancey JO, Klarskov P, Shull BL, Smith AR. The standardization of terminology of female pelvic organ prolapse and pelvic floor dysfunction. Am J Obstet Gynecol. 1996 Jul;175(1):10-7. doi: 10.1016/s0002-9378(96)70243-0. PMID 8694033